CLINICAL TRIAL: NCT02616055
Title: Long-Term Treatment and Follow up of Subjects Completing 24 Months of Treatment With Tesevatinib on Study KD019-101 in Subjects With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Long-Term Treatment and Follow up of Subjects Completing 24 Months of Treatment With Tesevatinib on Study KD019-101
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor opened Phase 2 Study.
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KD019-207
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — XL647

STUDY DESIGN:
Intervention Model Description: Extension Study, participants to be followed at the dose of tesevatinib they were receiving in Study KD019-101.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 50mg Daily (Experimental): One 50mg tesevatinib tablet per day
  Interventions: Drug: tesevatinib
- 100mg Daily (Experimental): Two 50mg tesevatinib tablets per day
  Interventions: Drug: tesevatinib
- 150mg M/Th (Experimental): Three 50mg tesevatinib tablets every Monday and Thursday.
  Interventions: Drug: tesevatinib
- 150mg MWF (Experimental): Three 50mg tesevatinib tablets every Monday, Wednesday and Friday.
  Interventions: Drug: tesevatinib

INTERVENTIONS:
Drug: tesevatinib
  Other Names: KD019; XL647

SUMMARY:
Subjects who received tesevatinib in Study KD019-101 and completed 24 months of treatment will continue on the dose of tesevatinib they were receiving at 24 months on the KD019-101 study.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have received 24 months of treatment with tesevatinib on study KD019-101. (Twenty-four months of study drug treatment includes days without treatment that were allowed by the KD019-101 protocol.)
* Sexually active subject (male and female) has agreed to use two forms of accepted methods of contraception during the course of the study and for 3 months after the last dose of study drug. Effective birth control includes (a) IUD plus one barrier method; (b) on stable doses of hormonal contraception for at least 3 months (eg, oral, injectable, implant, transdermal) plus one barrier method; or (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm).
* Female subjects of childbearing potential have a negative pregnancy test at screening. Females of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-12-25; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Monitor Longitudinal Changes in Estimated Glomerular Filtration Rate | 37 Months
  Monitor longitudinal changes in estimated glomerular filtration rate (eGFR) in subjects with ADPKD when treated with tesevatinib.

SECONDARY OUTCOMES:
Monitor Longitudinal Changes in Total Kidney Volume | 37 Months
  Monitor longitudinal changes from baseline in total kidney volume (TKV) in subjects with ADPKD when treated with tesevatinib.
Number of Subjects Experiencing Adverse Events as a Measure of Safety and Tolerability | 37 Months
  To evaluate the long term safety and tolerability of tesevatinib in subjects with ADPKD when treated with tesevatinib.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - University of Virginia - Nephrology Clinical Research Center, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin